CLINICAL TRIAL: NCT01336673
Title: An Observational Study on the Use of Glucophage XR® Therapy in the Management of Patients With Type 2 Diabetes
Brief Title: Glucophage XR® Observational Study
Status: Terminated | Type: Observational
Why Stopped: The study was scheduled for completion February 2013. Because of difficulties encountered in completing the trial the study was terminated by sponsor June 2013.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Ltd., Thailand (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR200039-503
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes Mellitus Type 2; GI Side Effect
Keywords: Glucophage XR; Tolerability
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a non-interventional, prospective study where no visits or additional interventions to the daily practice of the physician will be performed. Glucophage XR® has recently been available in Thailand for the treatment of patients with type 2 diabetes. A prospective observational study will be valuable to provide information on the day-to-day experience of using Glucophage XR® in the management of this patient population. The data may provide an insight into the use of Glucophage XR® in routine clinical practice in Thailand.

DETAILED DESCRIPTION:
Metformin (Glucophage) is the standard first line therapy for patients with type 2 diabetes mellitus. The landmark UK Prospective Diabetes Study Group demonstrated significant reduction in the risk of myocardial infarction and overall mortality in overweight patients with type 2 diabetes treated with metformin and metformin was more effective in controlling blood glucose compared with lifestyle only diet-based policy. The observed improvement of blood glucose was not associated with weight gain or hypoglycaemia in contrast to treatment with either a sulphonylurea or insulin.

It is well accepted that patients' compliance with therapy tends to decrease as the dosage frequency increases and that regimens should be simplified as far as possible to support good compliance with therapy. The use of an extended-release formulation of metformin (Glucophage XR®) may support the simplification of treatment for patients by allowing a once-daily administration of metformin.

Although patients taking metformin had significantly lower fasting and postprandial plasma glucose and hemoglobin A1C concentrations, they also had a higher prevalence of Gastrointestinal (GI) side effects. The most commonly reported symptoms was diarrhea (53,2 % compared to 11,7% on placebo). In a study employing self-administered questionnaires to ascertain GI symptoms in patients with type 2 diabetes approximately 20% of those taking immediate-release metformin reported diarrhea as the most common symptoms. Although less than 5% of patients discontinue metformin treatment for this reason, such adverse events can be troublesome, may limit the dosage of metformin and may impair compliance with therapy. Glucophage XR may lead to improved tolerability, by smoothing the peaks and troughs in metformin plasma concentrations and delaying the achievement of peak plasma concentration, compared with an immediate-release formulation. Initial placebo-controlled clinical trials with Glucophage XR indicate that 9,6% patients reported diarrhea (compare to 1,5% on placebo).

Thus, the use of Glucophage XR® may provide benefits in terms of improved patient management, by enabling once-daily dosing and reducing the incidence of gastrointestinal side effects for some patients. A prospective observational study will be valuable to provide information on the day-to-day experience of using Glucophage XR® in the management of this patient population. The data may provide an insight into the use of Glucophage XR® in routine clinical practice in Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 2 diabetes
* Considered as suitable for treatment Glucophage XR®
* Agreeing to maintain prior diet and exercise habits during the full course of the study
* Patient is regularly followed by/monitored by the investigator for type II diabetes mellitus
* Patients for whom a written informed consent has been obtained

Exclusion Criteria:

* Contraindicated use of Glucophage XR based on local label
* Renal disease or renal dysfunction
* Acute or chronic metabolic acidosis, including diabetic ketoacidosis, with or without coma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged > 18 and diagnosed with type 2 diabetes and considered by physician as suitable for treatment Glucophage XR®
Sampling Method: Non-Probability Sample
Enrollment: 518 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who experience at least one gastrointestinal side effect | 12 weeks

SECONDARY OUTCOMES:
Proportion of patients who discontinue Glucophage XR® prematurely, defined as less than 12 weeks, due to side effects. | 12 weeks
Incidence of side effects | 12 weeks
Change of Hemoglobin A1c level from baseline after at least 12 weeks of Glucophage XR® therapy | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research Manager, Study Director — Merck Ltd., Thailand, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Faculty of Medicine Vajira Hospital, Bangkok, Thailand